CLINICAL TRIAL: NCT04868006
Title: The Effect of End-range Maitland Mobilization on Glenohumeral Internal Rotation Deficit and Proprioception in Volleyball Players
Brief Title: End-range Maitland Mobilization on Glenohumeral Internal Rotation Deficit and Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Maitland_GIRD
Record Dates: First submitted 2021-04-22; First posted 2021-04-30 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Sports Physical Therapy
Keywords: Musculoskeletal Manipulations; Range Of Motion, Articular; Proprioception; Volleyball

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- End-range mobilization + proprioception training (Experimental): End-range Maitland mobilization performed in end-range internal rotation of the shoulder accompanied with 8--week long proprioception training
  Interventions: Procedure: End-range Maitland mobilization + proprioception training
- Non end-range mobilization+ proprioception training (Active Comparator): Non end-range Maitland mobilization performed in loose position of the shoulder accompanied with 8--week long proprioception training
  Interventions: Procedure: Non end-range Maitland mobilization + proprioception training
- Sham manual therapy technique + proprioception training (Sham Comparator): Placebo performed in loose position of the shoulder accompanied with 8--week long proprioception training
  Interventions: Procedure: Sham manual therapy technique + proprioception training

INTERVENTIONS:
Procedure: End-range Maitland mobilization + proprioception training — End-range Maitland mobilization performed in end position of internal rotation of the shoulder accompanied with 8--week long proprioception training
  Arms: End-range mobilization + proprioception training
Procedure: Non end-range Maitland mobilization + proprioception training — Non end-range Maitland mobilization performed in loose position of the shoulder accompanied with 8--week long proprioception training
  Arms: Non end-range mobilization+ proprioception training
Procedure: Sham manual therapy technique + proprioception training — Placebo performed in loose position of the shoulder accompanied with 8--week long proprioception training
  Arms: Sham manual therapy technique + proprioception training

SUMMARY:
Glenohumeral internal rotation deficit (GIRD) is one of the main reasons for glenohumeral pain in athletes with over-head activity. As GIRD increases, the ratio between internal and external rotation changes resulting in decreased joint stability.

Joint mobilization is a possible option for the decrease of GIRD and contribution to improvement of proprioception in addition to physical therapy. The aim of this trial is to investigate the effect of end-range Maitland mobilization in addition to physical therapy on GIRD, other joint movements and proprioception.

DETAILED DESCRIPTION:
Glenohumeral internal rotation deficit (GIRD) is one of the main reasons for glenohumeral pain in athletes with over-head activity. As GIRD increases, the ratio between internal and external rotation changes resulting in decreased joint stability. The occurence of GIRD and decreased joint proprioception may lead to different shoulder pathologies (e.g. Impingement syndrome).

Joint mobilization is a possible option for the decrease of GIRD and contribution to improvement of proprioception in addition to physical therapy. Several joint mobilization techniques exists, which can be applied for stretching of periarticular tissues. Maitland mobilization is a well applied mobilization type. The effectiveness of both end-range and not end-range Maitland mobilization in lengthening of periarticular tissues and improvement of joint proprioception has been previously confirmed amongst several diseases. However, the effect of end-range Maitland mobilization on decrease of GIRD and proprioception in addition to physical therapy has not been investigated in volleyball players so far.

The aim of this trial is to investigate the effect of end-range Maitland mobilization in addition to physical therapy on GIRD, other joint movements and proprioception.

ELIGIBILITY:
Inclusion Criteria:

* National Championship players in I. or II. level
* at least, 10 degree deficit of glenohumeral internal rotation in the dominant shoulder compared to the non-dominant hand

Exclusion Criteria:

* previous trauma or surgery on the dominant shoulder
* participation in any kind of treatment during the intervention period

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Internal rotation of the dominant glenohumeral joint | after 8 weeks
  Measurement of active internal rotation of the dominant glenohumeral joint with goniometer expressed in degree

SECONDARY OUTCOMES:
Flexion of the dominant glenohumeral joint | after 8 weeks
  Measurement of active flexion of the dominant glenohumeral joint with goniometer expressed in degree
Extension of the dominant glenohumeral joint | after 8 weeks
  Measurement of active extension of the dominant glenohumeral joint with goniometer expressed in degree
Abduction of the dominant glenohumeral joint | after 8 weeks
  Measurement of active abduction of the dominant glenohumeral joint with goniometer expressed in degree
Adduction of the dominant glenohumeral joint | after 8 weeks
  Measurement of active adduction of the dominant glenohumeral joint with goniometer expressed in degree
External rotation of the dominant glenohumeral joint | after 8 weeks
  Measurement of active external rotation of the dominant glenohumeral joint with goniometer expressed in degree
Western Ontario Shoulder Instability Index | after 8 weeks
  Western Ontario Shoulder Instability Index of the dominant shoulder
Posterior Shoulder Endurance Test | after 8 weeks
  Muscle strength test of the dominant shoulder expressed in Newton
Proprioception of the shoulder | after 8 weeks
  Proprioception of the shoulder measured with plurimeter expressed in degree
Davies test | after 8 weeks
  Measurement of proprioception and muscle strength test by the Davies test expressed in amount of success touch
Sportspecific proprioception test | after 8 weeks
  Measurement of the precision of serving expressed in centimeter

CONTACTS AND LOCATIONS:
Overall Officials: Miklós Pozsgai, Principal Investigator — Harkány Thermal Rehabilitation Centre
Locations (1):
- Harkány Thermal Rehabilitation Centre, Harkány, Please Select, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Miura K, Tsuda E, Ishibashi Y. Glenohumeral Rotational Deficit and Suprascapular Neuropathy in the Hitting Shoulder in Male Collegiate Volleyball Players. Prog Rehabil Med. 2019 Jan 12;4:20190002. doi: 10.2490/prm.20190002. eCollection 2019. PMID 32789249
- [Result] Wilk KE, Reinold MM, Macrina LC, Porterfield R, Devine KM, Suarez K, Andrews JR. Glenohumeral internal rotation measurements differ depending on stabilization techniques. Sports Health. 2009 Mar;1(2):131-6. doi: 10.1177/1941738108331201. PMID 23015864